CLINICAL TRIAL: NCT06248853
Title: Effect of Graston Technique on Planter Thickness in Patients With Planter Fasciitis
Acronym: PF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator nabil mahmoud ismail abdel-aal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002947
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fascitis
Keywords: graston technique; planter thickness; planter fasciitis
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Graston technique and exercise program
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Garston technique (Experimental): the patients will receive graston technique with exercise program three times aweek for six weeks
  Interventions: Other: Garston technique; Other: exercise program
- exercise program (Active Comparator): the patients will receive an exercise program three times a week for six weeks
  Interventions: Other: exercise program

INTERVENTIONS:
Other: Garston technique — the patients will receive instrumented assisted soft tissue mobilization using the Graston technique, which includes the application of a cream to the posterior calf and plantar foot from the knee to the toes to reduce friction on the skin. The Graston tools will be used to mobilize the tissues of the triceps surae and plantar foot bypassing the tools along the leg and foot
  Arms: Garston technique
Other: exercise program — the patients will receive pedaling an exercise bicycle for 5 min with minimal resistance to warm the tissues, gastrocnemius stretches performed on a step for three repetitions held for 30 sec each , plantar fascia stretching performed in a seated position for three repetitions held for 30 sec each, and foot intrinsic muscular strengthening using a short foot exercise. Ice will be offered as needed for pain management after each session in addition to home program exercise

SUMMARY:
this study will be conducted to investigate the effect of Graston Technique on Planter Thickness in Patients With Planter Fasciitis

DETAILED DESCRIPTION:
Plantar fasciitis (PF), generally a self-limiting condition, is identified as one of the most common causes of heel pain in adults. It affects both sedentary and athletic populations .

It may be considered that PF emerges due to excessive and prolonged standing or running, which causes an acute inflammation or micro-tears, and degenerative changes plantar fascia. The persistence of these risk factors inhibits the regular repair process thus collagen degeneration occurs, causing the structural changes of the plantar fascia. Numerous interventions have been described for treatment of PF, which include: Stretching calf or plantar region which is performed with the patient stands with staggered legs facing toward a wall, with both hands stretched out .The Graston technique can break up scar tissue and restore soft tissue. The Graston technique is a type of manual therapy in which patented stainless-steel instruments are used to restore soft tissue motion by breaking up scar tissue. fifty patients with planter fasciitis will be assigned randomly to two equal groups; first one will receive graston technique in addition to exercise program, the second one will receive exercise program only for six weeks

ELIGIBILITY:
Inclusion Criteria:

* patients that Clinically diagnosed cases of plantar fasciitis not less than 6 weeks.
* patients willing to precipitate in the study and take treatment for 6 successive weeks.
* Heel pain felt maximally over the plantar aspect of heel
* Pain in the heel on the first step in the morning
* No history of rest pain in the heel

Exclusion Criteria:

* Subjects with clinical disorders where therapeutic ultrasound is contraindicated such as infective conditions of foot, tumor, calcaneal fracture, metal implant around ankle.
* Subjects with a clinical disorder where myofascial release is contraindicated as dermatitis.
* Subjects with impaired circulation to lower extremities
* Subjects with referred pain due to sciatica and other neurological disorders.
* Arthritis
* Corticosteroids injection in heel preceding 3 months

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
plantar thickness | up to six weeks
  Ultrasonography will be used to measure planter thickness

SECONDARY OUTCOMES:
pain intensity | up to six weeks
  Visual Analogue Scale (VAS) will be used to assess pain intensity: The VAS is a 100-mm horizontal line that may be used to quantify symptoms in a continuous fashion. Patients will instructed to indicate the intensity of their pain by marking on a line anchored by "no pain" on the left and "worst imaginable pain" on the right .
pain intensity at the first step | up to six weeks
  numerical pain rating scale (NPRS) will be used to measure pain intensity at the first step. NPRS is a 10cm horizontal line t. Patients will instructed to indicate the intensity of their pain by marking on a line anchored by "no pain" on the left and "worst imaginable pain" on the right side.
functional levels of foot | up to six weeks
  The Foot and Ankle Ability Measure (FAAM) questionnaire will be used to assess foot function. The FAAM is a self-reported questionnaire that comprehensively assesses the physical function of those with musculoskeletal conditions of the leg, foot, and ankle. It has a 21-item subscale for measuring the function of the individual with his or her activities of daily living (ADLs) and a ten-item subscale for measuring function with sports. The ADL subscale will be used for this study. The instrument is scored on a Likert scale from 4 to 0, with 4 representing ''no difficulty'' as going up stairs and 0 representing ''unable to do.'' The answers are then converted to a scale from 0 to 100, with a higher score representing a higher functional level.
pain pressure threshold | up to six weeks
  The pressure algometer device will be used to measure pain pressure threshold